CLINICAL TRIAL: NCT05940389
Title: Nasolabial Soft Tissue Esthetics and Maxillary Changes in Unilateral Cleft Lip and Palate Using PreSurgical Infant Orthopedics With Different Approaches: A Parallel-arm Randomized Clinical Trial
Brief Title: Nasolabial Soft Tissue Esthetics and Maxillary Changes in Unilateral Cleft Lip and Palate Using PreSurgical Infant Orthopedics With Different Approaches
Acronym: PSIO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Al-Azhar University (Other)
Collaborators: Innovinity medical hub (Unknown); Smile train (Unknown)
Responsible Party: Principal Investigator, Abdallah Mohammad Baha El-Din Mohammed, Assistant lecturer, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Innovinity Medical Hub
Record Dates: First submitted 2023-06-23; First posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Unilateral Cleft Lip; Nasoalveolar Molding
Keywords: NAM; UCLP; pre-surgical orthopedics; DynaCleft

STUDY DESIGN:
Intervention Model Description: A randomized clinical trial, parallel arm, superiority framework with 1:1 allocation ratio.
Who Masked: Outcomes Assessor
Masking Description: The study will be single-blinded. The outcome assessors will be blinded as the measurements will be done on laser-scanned casts and 3D facial images. The operator and the patient's parent cannot be blinded due to the nature of the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NAM appliance Group (Experimental): The NAM appliance is constructed according to the Grayson technique [8] with the nasal stent added from the start. The adhesive paste is used to hold the alveolar plate in place and labial taping is used. Patients are followed each 2 to 3 weeks for the appliance to be relined and selectively ground to modify the pressure as needed. The surgical lip repair technique involved will be done by one surgeon using the Delare technique without the blind dissection of the alar cartilage.
  Interventions: Device: Naso Alveolar Mold
- Taping with nasal elevator: (Experimental): For the lip approximation, Airoplast tape is used which is water resistant transparent and coated with hypoallergic adhesive on one side. The nasal elevator is 3D printed from the design inspired by the Dynacleft nasal elevator. Patients will be followed each 2 to 3 weeks for any modifications or adjustments.
  The surgical lip repair technique involved will be done by one surgeon using the Delare technique without the blind dissection of the alar cartilage.
  Interventions: Device: Taping with nasal elevator:

INTERVENTIONS:
Device: Naso Alveolar Mold — The NAM appliance is constructed according to the Grayson technique [8] with the nasal stent added from the start. The adhesive paste is used to hold the alveolar plate in place and labial taping is used. Patients are followed each 2 to 3 weeks for the appliance to be relined and selectively ground to modify the pressure as needed.
  Other Names: NAM
  Arms: NAM appliance Group
Device: Taping with nasal elevator: — For the lip approximation, Airoplast tape is used which is water resistant transparent and coated with hypoallergic adhesive on one side. The nasal elevator is 3D printed from the design inspired by the Dynacleft nasal elevator. Patients will be followed each 2 to 3 weeks for any modifications or adjustments.
  Other Names: DYNA
  Arms: Taping with nasal elevator:

SUMMARY:
The nasal deformity is an abnormality in the appearance and structure of the nose in cleft patients having unilateral cleft lip and palate (UCLP). It involves the displacement of the lower lateral nasal cartilage, oblique and short columella, depressed dome, overhanging nostril apex, and deviated septum. Difficulty in breathing and smelling are the main problems of this deformity. Rhinoplasty for CLP patients is very complicated due to the complex nature of this type of deformity, especially in wide and bilateral cleft patients it is quite challenging.

DETAILED DESCRIPTION:
The nasal deformity is an abnormality in the appearance and structure of the nose in cleft patients having unilateral cleft lip and palate (UCLP). It involves the displacement of the lower lateral nasal cartilage, oblique and short columella, depressed dome, overhanging nostril apex, and deviated septum. Difficulty in breathing and smelling are the main problems of this deformity. Rhinoplasty for CLP patients is very complicated due to the complex nature of this type of deformity, especially in wide and bilateral cleft patients it is quite challenging. The cleft width along with the nasal deformity and collapse in the nasal cartilage could affect the outcome of the surgical lip closure with the cleft width as a major factor affecting the tension produced in the closure and future collapse of the nose. There is a striking diversity in the literature regarding treatment protocols for UCLP, with no standardized management protocols . Clinical decision-making based on evidence is lacking due to the few randomized clinical trials comparing the effectiveness of different approaches. A recent systematic review conducted a comprehensive search aiming at identifying the different treatment protocols and effectiveness of using pre-surgical infant orthopedics (PSIO) and recommended the need for further well-designed and high-quality randomized clinical trials (RCTs) in this area due to the unstandardized protocols with high diversity. Various studies supported the positive effect of naso-alveolar molding (NAM) appliance therapy on nasal symmetry in UCLP treatment. The NAM therapy decreases the severity of the initial cleft deformity and repositions deformed nasal cartilage and alveolar process, which has many beneficial results in the surgery outcome. Taping has been assessed in infants with UCLP and was deemed successful as well by a few studies. To our knowledge, no RCTs are comparing the use of NAM therapy to taping with the use of nasal elevators on UCLP patients.

ELIGIBILITY:
Inclusion Criteria:

* Infants with 0 (after birth) to 1 month of age
* Non-syndromic with no other medical conditions
* Unilateral complete cleft lip and palate
* Cleft width > 5 mm

Exclusion Criteria:

* Syndromic UCLP or bilateral cleft lip and palate
* Incomplete UCLP
* Cleft width ≤ 5 mm

Ages: 1 Day to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in nasal tip projection | T0= before Intervention, T1=immediately before surgery, T2 1 month after surgery, T3= 6 months after surgery, T4= 1 year after surgery
  Observing the change in the nasolabial angle by the superimposition of the 3D facial scans at different time points (T0, T1, T2, T3, and T4)
change in Columella height | T0= before Intervention, T1=immediately before surgery, T2 1 month after surgery, T3= 6 months after surgery, T4= 1 year after surgery
  observing the change in the linear distance (mm) from the subnasal point to the labral superiors point by the superimposition of the 3D facial scans at different time points (T0, T1, T2,T3, and T4)
Change in projection alar length | T0= before Intervention, T1=immediately before surgery, T2 1 month after surgery, T3= 6 months after surgery, T4= 1 year after surgery
  Observing the change in the linear distance (mm) from the most anterior point of the affected nasal ala to the deepest point at the base of the nose by the superimposition of the 3D facial scans at different time points (T0, T1, T2, T3, and T4)
Change in width of the nostril | T0= before Intervention, T1=immediately before surgery, T2 1 month after surgery, T3= 6 months after surgery, T4= 1 year after surgery
  Observing the change in the linear distance (mm) from the most lateral point of the affected nasal ala to the most medial point of the affected ala by the superimposition of the 3D facial scans at different time points (T0, T1, T2, T3, and T4)
Change in nasal basal width | T0= before Intervention, T1=immediately before surgery, T2 1 month after surgery, T3= 6 months after surgery, T4= 1 year after surgery
  Observing the change in the linear distance (mm) from the most lateral point of the affected nasal ala to the most medial point of the affected ala at the level of the nasal base by the superimposition of the 3D facial scans at different time points (T0, T1, T2, T3, and T4)
Change in the angle of the columella | T0= before Intervention, T1=immediately before surgery, T2 1 month after surgery, T3= 6 months after surgery, T4= 1 year after surgery
  Observing the change in the columella-labial angle by the superimposition of the 3D facial scans at different time points (T0, T1, T2, T3, and T4)
Change in cleft lip segment | T0= before Intervention, T1=immediately before surgery, T2 1 month after surgery, T3= 6 months after surgery, T4= 1 year after surgery
  Observing the change in the width (mm) of the labial cleft segment from the most lateral point to the most medial point at the widest area of the labial cleft by the superimposition of the 3D facial scans at different time points (T0, T1, T2, T3, and T4)
Change in the height of the non-cleft lip | T0= before Intervention, T1=immediately before surgery, T2 1 month after surgery, T3= 6 months after surgery, T4= 1 year after surgery
  Observing the change in the non-affected lip height (mm) from the subnasal point to the labral superior point by the superimposition of the 3D facial scans at different time points (T0, T1, T2, T3, and T4)
Change in the height of the cleft lip | T0= before Intervention, T1=immediately before surgery, T2 1 month after surgery, T3= 6 months after surgery, T4= 1 year after surgery
  Observing the change in the affected lip height (mm) from the subnasal point to the labral superior point by the superimposition of the 3D facial scans at different time points (T0, T1, T2, T3, and T4)

SECONDARY OUTCOMES:
Change in the alveolar cleft width | T0= before Intervention, T1=immediately before surgery, T2 1 month after surgery, T3= 6 months after surgery, T4= 1 year after surgery
  Observing the change in the alveolar cleft width (mm) from the most lateral to the most medial points at cleft edges by the superimposition of the 3D occlusal scans at different time points (T0, T1, T2, T3, and T4)
Change in arch perimeter | T0= before Intervention, T1=immediately before surgery, T2 1 month after surgery, T3= 6 months after surgery, T4= 1 year after surgery
  Observing the change in the arch perimeter (mm) from the most left and right posterior points by the superimposition of the 3D occlusal scans at different time points (T0, T1, T2, T3, and T4)
Change in greater segment perimeter | T0= before Intervention, T1= after 1 month, T2= after 6 months, T3=after 1 year
  observing the change in the greater segment perimeter (mm) from the most posterior point to the most anterior point at the cleft edge by the superimposition of the 3D occlusal scans at different time points (T0, T1, T2, T3, and T4)
Change in lesser segment perimeter | T0= before Intervention, T1=immediately before surgery, T2 1 month after surgery, T3= 6 months after surgery, T4= 1 year after surgery
  observing the change in the lesser segment perimeter (mm) from the most posterior point to the most anterior point at the cleft edge by the superimposition of the 3D occlusal scans at different time points (T0, T1, T2, T3, and T4)
Change in posterior width of the palatal cleft | T0= before Intervention, T1=immediately before surgery, T2 1 month after surgery, T3= 6 months after surgery, T4= 1 year after surgery
  observing the change in the posterior cleft width (mm) at the primary molars' gum pads by the superimposition of the 3D occlusal scans at different time points (T0, T1, T2, T3, and T4)
Change in arch width at the anterior region | T0= before Intervention, T1=immediately before surgery, T2 1 month after surgery, T3= 6 months after surgery, T4= 1 year after surgery
  observing the change in the anterior arch width (mm) at the primary canine gum pads by the superimposition of the 3D occlusal scans at different time points (T0, T1, T2, T3, and T4)
Change in greater segment rotation | T0= before Intervention, T1=immediately before surgery, T2 1 month after surgery, T3= 6 months after surgery, T4= 1 year after surgery
  observing the change in the angle between the greater segment and midsagittal plane by the superimposition of the 3D occlusal scans at different time points (T0, T1, T2,T3 and T4)
Change in lesser segment rotation | T0= before Intervention, T1=immediately before surgery, T2 1 month after surgery, T3= 6 months after surgery, T4= 1 year after surgery
  observing the change in the angle between the lesser segment and midsagittal plane by the superimposition of the 3D occlusal scans at different time points (T0, T1, T2, T3, and T4)
Change in arch width at the posterior region | T0= before Intervention, T1=immediately before surgery, T2 1 month after surgery, T3= 6 months after surgery, T4= 1 year after surgery
  observing the change in the posterior arch width (mm) at the primary molars' gum pads by the superimposition of the 3D occlusal scans at different time points (T0, T1, T2, T3, and T4)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Padovano WM, Skolnick GB, Naidoo SD, Snyder-Warwick AK, Patel KB. Long-Term Effects of Nasoalveolar Molding in Patients With Unilateral Cleft Lip and Palate: A Systematic Review and Meta-Analysis. Cleft Palate Craniofac J. 2022 Apr;59(4):462-474. doi: 10.1177/10556656211009702. Epub 2021 Apr 22. PMID 33882703
- [Background] Wadde K, Chowdhar A, Venkatakrishnan L, Ghodake M, Sachdev SS, Chhapane A. Protocols in the management of cleft lip and palate: A systematic review. J Stomatol Oral Maxillofac Surg. 2023 Apr;124(2):101338. doi: 10.1016/j.jormas.2022.11.014. Epub 2022 Nov 21. PMID 36410660
- [Background] Saad MS, Fata M, Farouk A, Habib AMA, Gad M, Tayel MB, Marei MK. Early Progressive Maxillary Changes with Nasoalveolar Molding: Randomized Controlled Clinical Trial. JDR Clin Trans Res. 2020 Oct;5(4):319-331. doi: 10.1177/2380084419887336. Epub 2019 Dec 20. PMID 31860800
- [Background] Abd El-Ghafour M, Aboulhassan MA, Fayed MMS, El-Beialy AR, Eid FHK, Hegab SE, El-Gendi M, Emara D. Effectiveness of a Novel 3D-Printed Nasoalveolar Molding Appliance (D-NAM) on Improving the Maxillary Arch Dimensions in Unilateral Cleft Lip and Palate Infants: A Randomized Controlled Trial. Cleft Palate Craniofac J. 2020 Dec;57(12):1370-1381. doi: 10.1177/1055665620954321. Epub 2020 Sep 10. PMID 32909815
- [Background] Chang CS, Wallace CG, Pai BC, Chiu YT, Hsieh YJ, Chen IJ, Liao YF, Liou EJ, Chen PK. Comparison of two nasoalveolar molding techniques in unilateral complete cleft lip patients: a randomized, prospective, single-blind trial to compare nasal outcomes. Plast Reconstr Surg. 2014 Aug;134(2):275-282. doi: 10.1097/PRS.0000000000000361. PMID 24732649
- [Background] Abd El-Ghafour M, Aboulhassan MA, El-Beialy AR, Fayed MMS, Eid FHK, El-Gendi M, Emara D. Is Taping Alone an Efficient Presurgical Infant Orthopedic Approach in Infants With Unilateral Cleft Lip and Palate? A Randomized Controlled Trial. Cleft Palate Craniofac J. 2020 Dec;57(12):1382-1391. doi: 10.1177/1055665620944757. Epub 2020 Aug 10. PMID 32772701
- [Background] Abd El-Ghafour M, Aboulhassan MA, El-Beialy AR, Fayed MMS, Eid FHK, Emara D, El-Gendi M. Does Presurgical Taping Change Nose and Lip Aesthetics in Infants with Unilateral Cleft Lip and Palate? A Randomized Controlled Trial. Plast Reconstr Surg. 2022 Dec 1;150(6):1300e-1313e. doi: 10.1097/PRS.0000000000009738. Epub 2022 Sep 20. PMID 36126199
- [Background] Grayson BH, Santiago PE, Brecht LE, Cutting CB. Presurgical nasoalveolar molding in infants with cleft lip and palate. Cleft Palate Craniofac J. 1999 Nov;36(6):486-98. doi: 10.1597/1545-1569_1999_036_0486_pnmiiw_2.3.co_2. PMID 10574667
- [Background] Castillo T, Luisa PPM, Clark P, Robertson JP, Montalva FM, Figueroa AA, Mejia ML, Moreno AS, Martinez MD, Aguilera A, Arreguin JC, Dosal MRP, de la Paz Aguilar Saavedra M, Granados A. Developing a core outcome set for anthropometric evaluation for presurgical infant orthopaedics for unilateral cleft lip and palate: e-Delphi consensus. J Plast Reconstr Aesthet Surg. 2022 Oct;75(10):3795-3803. doi: 10.1016/j.bjps.2022.06.065. Epub 2022 Jun 24. PMID 36075806
- [Background] Yu Q, Gong X, Shen G. CAD presurgical nasoalveolar molding effects on the maxillary morphology in infants with UCLP. Oral Surg Oral Med Oral Pathol Oral Radiol. 2013 Oct;116(4):418-26. doi: 10.1016/j.oooo.2013.06.032. PMID 24035109
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343